CLINICAL TRIAL: NCT07249658
Title: Effects of Power and High-Intensity Gait Training for Functional Mobility an Ambulation in Chronic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02166 / Fatima Khan
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Stroke
Keywords: gait training; strength; power; functional mobility; ambulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: power training + high-intensity gait training (Experimental): This group will be given a combined program that comprises gait training and lower-limb power training, three times a week. The gait component will consist of overground walking at increased intensity and treadmill training whilst using a safety harness. At the initial stage, treadmill (1.5-2.0 mph) for a duration of 2 sets,3 minutes, and 10-minute overground moderate-intensity walking is offered with frequent rests. The intensity will be gradually increased throughout the program, with an increase in speeds on the treadmill to 2.0 mph (2.5 mph or 3.0 mph) (two sets of three minutes, then three sets of 3-4 minutes, and finally 5-10 minutes at moderate and high intensity) and overground walking (10-15 min to up to 20 min at high intensity).
  Interventions: Other: power training + high-intensity gait training
- Control 1: power training (Active Comparator): Individuals in the power training group will also train three times a week, including lower-limb resistance and functional strength work, applying a focus on explosive concentric effort. The exercise will consist of 3 sets (or 6 repetitions of stepping backward over a hurdle, warming up in sitting knee extension with resistance band, marching in a seat with a load on the ankle, transferring sit to stand, and hopping up on the box 46 inch). The number of sets will be increased as they are tolerated, beginning with 3 sets to 4 sets and ultimately up to 5 sets of each exercise as tolerated as the training progresses. The intensity will be progressed by raising the resistance ( box height) and performance speed.
  Interventions: Other: power training
- Control 2: High-intensity gait training (Active Comparator): This group will receive high-intensity gait training three days per week, taking into consideration both treadmill gait in a safety harness and overground gait. Initial training will start with a treadmill speed of 1.5 2.0 mph, two sets/3 minutes each, and 15 minutes overground walking at moderate intensity, and rest breaks when necessary. The progression will entail a gradual increase in the speeds on the treadmill to 2.0-2.5 mph (three sets of 3 minutes) and subsequently to 2.5 3.0 mph (three sets of 3 4 minutes) with the overground walking time extended to 15-20 mins and subsequently to 20 minutes at greater intensities.
  Interventions: Other: high-intensity gait training

INTERVENTIONS:
Other: power training + high-intensity gait training — This group will be given a combined program that comprises gait training and lower-limb power training, which will take place three times a week. The gait component will consist of overground walking at increased intensity and treadmill training whilst using a safety harness. At the initial stage, treadmill (1.5-2.0 mph) for a duration of 2 sets,3 minutes, and 10-minute overground moderate-intensity walking is offered with frequent rests. The intensity will be gradually increased throughout the program, with an increase in speeds on the treadmill to 2.0 mph (2.5 mph or 3.0 mph) (two sets of three minutes, then three sets of 3-4 minutes, and finally 5-10 minutes at moderate and high intensity) and overground walking (10-15 min to up to 20 min at high intensity).
  Arms: Experimental: power training + high-intensity gait training
Other: power training — Individuals in the power training group will also train three times a week, including lower-limb resistance and functional strength work, applying a focus on explosive concentric effort. The exercise will consist of 3 sets (or 6 repetitions of stepping backward over a hurdle, warming up in sitting knee extension with resistance band, marching in a seat with a load on the ankle, transferring sit to stand, and hopping up on the box 46 inch). The number of sets will be increased as they are tolerated, beginning with 3 sets to 4 sets and ultimately up to 5 sets of each exercise as tolerated as the training progresses. The intensity will be progressed by raising the resistance ( box height) and performance speed.
  Arms: Control 1: power training
Other: high-intensity gait training — The members of this group will receive high-intensity gait training three days per week, taking into consideration both treadmill gait in a safety harness and overground gait. Initial training will start with a treadmill speed of 1.5 2.0 mph, two sets/3 minutes each, and 15 minutes overground walking at moderate intensity, and rest breaks when necessary. The progression will entail a gradual increase in the speeds on the treadmill to 2.0-2.5 mph (three sets of 3 minutes) and subsequently to 2.5 3.0 mph (three sets of 3 4 minutes) with the overground walking time extended to 15-20 mins and subsequently to 20 minutes at greater intensities.
  Arms: Control 2: High-intensity gait training

SUMMARY:
This randomized controlled trial aims to determine the combined effect of power training and high-intensity gait training on functional mobility and locomotion following chronic stroke.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of long-term disability, leaving many survivors with persistent motor and gait impairments such as muscle weakness, poor coordination, stiffness, and balance deficits. These problems often manifest as trunk and pelvic asymmetry, postural imbalance, and impaired weight shifting, resulting in abnormal gait patterns and reduced independence in daily life. Such limitations highlight the urgent need for effective, evidence-based rehabilitation strategies.

Power training, which emphasizes high-velocity resistance exercises, has been shown to enhance torque development in the paretic limb and improve walking speed, endurance, and spatiotemporal gait parameters in chronic stroke survivors. Similarly, high-intensity gait training (HIGT), which involves repetitive walking at challenging intensities, has demonstrated improvements in gait quality, endurance, and lower-limb biomechanics, particularly when integrated with robotic exosuits or structured clinical protocols. Both interventions have proven effective in enhancing functional mobility and quality of life.

However, research on the combined effects of power training and HIGT remains limited. This study aims to address this gap by examining how their synergistic application can optimize locomotion, reduce long-term disability, and promote social reintegration in individuals with chronic stroke. By providing evidence for more effective rehabilitation protocols, the findings have the potential to improve patient outcomes, reduce healthcare costs, and advance clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age
* more than ≥6 months of stroke onset
* first-ever unilateral ischemic stroke
* walking 10 meters independently with or without an assistive device
* being an independent ambulator (Functional Ambulation category >3)

Exclusion Criteria:

* people with a history of mental/cognitive illness
* combination with peripheral neuropathy
* having resting blood pressure above 160/100 mmHg even after taking medications;
* hemorrhagic stroke
* cardiovascular comorbidity
* any musculoskeletal condition that prevents or limits the participants from doing resistance training

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-02-21 (Estimated); Study Completion 2026-02-21 (Estimated)

PRIMARY OUTCOMES:
five times sit-to-stand test (FTSST) | 6 weeks
  The FTSST developed by Csuka and McCarty (1985) is a very reliable tool to measure sitting and standing performance as well as lower limb muscle strength and balance. It is a single-item test where the participant is required to rise from a chair and sit down five consecutive times as quickly as possible without using the arms. The score is recorded as the total time taken in seconds to complete the task.
Tmed Up and Go Test | 6 weeks
  The Timed Up and Go (TUG) is a commonly used outcome measure that can assess activity limitations in the ICF model by examining the patient's ability to ambulate and perform transfers.
10 meter Walk Test | 6 weeks
  The 10-Meter Walk Test was developed as a simple, quick, and reliable measure of gait speed. It is a single-item test where the participant walks 10 meters, with timing recorded for the middle 6 meters to exclude acceleration and deceleration phases. It is widely used to assess functional mobility, walking ability, and community ambulation in populations such as stroke, Parkinson's disease, geriatrics, and rehabilitation patients.
Barthel index | 6 weeks
  Assesses the level of independence in daily activities, such as feeding, bathing, and mobility, in individuals with physical disabilities. Literature showed strong criterion-related validity against the BI, with high reliability. This scoring system may become a convenient tool, allowing anyone to assess ADL.
Functional Gait Assessment | 6 weeks
  Measures balance and gait under various challenging conditions to assess fall risk and overall gait stability. The Functional Gait Assessment is a reliable, valid tool. It is composed of 10 items, each scored 0-3 (0 = severe impairment, 3 = normal performance). Maximum score = 30. Lower scores indicate higher risk of falls; ≤22/30 is often used as a cutoff for increased fall risk.

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Khan, MS-NMPT*, Principal Investigator — Riphah International Unversity; Arshad Nawaz Malik, PhD Rehab, Study Chair — Riphah International Unversity
Locations (1):
- National institute of Rehabilitation Medicine, NIRM, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No